CLINICAL TRIAL: NCT05313282
Title: A Randomized Controlled, Open-label, Multicenter Phase III Clinical Trial to Evaluate the Effectiveness and Safety of Hepatic Arterial Infusion Chemotherapy (HAIC) of Oxaliplatin, 5-fluorouracil and Leucovorin (mFOLFOX7) Combined With Apatinib and Camrelizumab Versus Apatinib and Camrelizumab for C-staged Hepatocellular Carcinoma in BCLC Classification.
Brief Title: A Trial of Hepatic Arterial Infusion Combined With Apatinib and Camrelizumab Versus Apatinib and Camrelizumab for C-staged Hepatocellular Carcinoma in BCLC Classification
Acronym: TRIPLET-III
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yang-kui Gu, Associate Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIPLET-III
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: C-staged Hepatocellular Carcinoma in BCLC Classification
Keywords: C-staged Hepatocellular Carcinoma; hepatic arterial infusion chemotherapy; anti-PD-1 immunotherapy; Camrelizumab; anti-angiogenic targeted therapy; Apatinib
MeSH Terms: interventions — apatinib; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): combination of hepatic arterial infusion chemotherapy (HAIC) of oxaliplatin, 5-fluorouracil and leucovorin (mFOLFOX7) , targeted drugs (Apatinib 250mg), and anti-PD-1 immunotherapy (Camrelizumab 200mg)
  Interventions: Combination Product: Hepatic Arterial Infusion combined with Apatinib and Camrelizumab
- control group (Active Comparator): combination of targeted drugs (Apatinib 250mg), and anti-PD-1 immunotherapy (Camrelizumab 200mg)
  Interventions: Combination Product: Apatinib combined with Camrelizumab

INTERVENTIONS:
Combination Product: Hepatic Arterial Infusion combined with Apatinib and Camrelizumab — Drug: FOLFOX Protocol (Oxaliplatin, fluorouracil, and leucovorin); Camrelizumab for injection and Apatinib-Mesylate Tablets Procedure: 1. On the first day of treatment, HAIC was conducted through a catheter intubated into the tumor feeding artery under DSA guidance with the following chemotherapeutic drugs (mFOLFOX7, oxaliplatin 85 mg/m2 2 hours, folinic acid 400 mg/m2, 5-FU 2500 mg/m2 46 hours) pumped into the tumor artery. The HAIC is repeated every 3 weeks. The cumulative maximum sessions of HAIC is up to 6 times.
  2. Taking Apatinib-Mesylate Tablets (250 mg/tablet) orally on the 8th day 30minutes after meals, once a day, for continuous medication.
  3. On the 22nd day of treatment, namely the second session of HAIC, intravenous infusion of Camrelizumab 200mg every 3 weeks.
  4. The cumulative maximum drug use period is up to 2 years. The patient is concurrent on medication until the treatment discontinuation criteria specified in the protocol appear.
  Arms: treatment group
Combination Product: Apatinib combined with Camrelizumab — Drug: Camrelizumab for injection and Apatinib-Mesylate Tablets Procedure: 1. Taking Apatinib-Mesylate Tablets (250 mg/tablet) orally 30minutes after meals, once a day, for continuous medication 2. Intravenous infusion of Camrelizumab 200mg every 2 weeks.
  Arms: control group

SUMMARY:
This study was designed to evaluate the effectiveness and safety of hepatic arterial infusion chemotherapy combined with Apatinib and Camrelizumab (treatment group) versus Apatinib and Camrelizumab (control group) for C-staged Hepatocellular Carcinoma in BCLC classification.

The primary outcome measure is to evaluate the progression-free-survival (PFS) of treatment group and control group for C-staged Hepatocellular Carcinoma in BCLC classification.

The secondary Outcome measures include the overall survival (OS), time to progress (TTP), time-to-response (TTR), duration of response (DOR), objective response rate (ORR) and disease control rate (DCR) of treatment group and control group for C-staged Hepatocellular Carcinoma in BCLC classification.

Moreover, this study aims to assess the safety and tolerability of treatment group and control group for C-staged Hepatocellular Carcinoma in BCLC classification.

DETAILED DESCRIPTION:
Primary liver cancer is a common malignant tumor of the digestive system in the world. There are about 854,000 new incidences and 810,000 mortality each year. In China, there is a high incidence of liver cancer, with about 466,000 new cases and 422,000 mortality each year. Hepatocellular carcinoma (HCC) accounted for about 90% of primary liver cancer in pathological type. Most patients have reached advanced stage or with distant metastasis when diagnosed and the natural median survival time is only 3 to 4 months. Then only systemic therapy is recommended for patients in advanced HCC in many global guidelines.

Hepatic arterial infusion chemotherapy (HAIC) of mFOLFOX7, anti-angiogenic targeting drugs, and antibody immunotherapy against programmed death molecule-1 (PD-1) immunological checkpoints are effective treatment options for advanced hepatocellular carcinoma. Many clinical studies have shown that the two-two combination of the above three treatment options can improve the anti-tumor overall response rate, the survival rate and even achieve clinical complete remission of patients with advanced HCC.

Shi Ming et al reported HAIC combined with systemic targeted therapy has a better survival outcome compared to systemic targeted therapy mono-therapy [OS 13.37 vs 7.13 months, PFS 7.03 vs 2.6 months] in JAMA Oncology. Although the toxicity of combination therapy is slightly higher than that of sorafenib monotherapy, these adverse effects are tolerable.

In addition, in a phase Ib study of Camrelizumab combined with apatinib in the treatment of advanced liver cancer, gastric cancer or gastroesophageal junction cancer showed that in 16 patients with HCC, the ORR was 50.0% and the DCR was 93.8%. When the dose of apatinib was 250 mg, the median PFS was 7.2 months. Camrelizumab combined with low dose apatinib can effectively reduce the incidence of adverse reactions, ≥10% of patients have treatment-related adverse reactions (all levels), no treatment-related adverse reactions leading to death. Therefore, low-dose anti-angiogenic drugs can inhibit tumor angiogenesis on the one hand, reduce immunosuppression by inducing normalization of blood vessels, enhance effector immune cell infiltration, and enhance anti-tumor immunity.

In summary, for patients of C-staged Hepatocellular Carcinoma, HAIC, anti-angiogenic targeted therapy, and anti-PD-1 immunotherapy have their important status, and the combination of any two treatments brings about synergy effect. Then, could the combination of the three treatment methods further improve the outcome of advanced hepatocellular carcinoma? A phase-II study conducted by our team revealed that a combination of hepatic arterial infusion chemotherapy, targeted drugs (Apatinib), and anti-PD-1 immunotherapy (Camrelizumab) showed promising clinical benefits and acceptable safety for BCLC Stage C HCC, as the confirmed ORR was 61.54% per RECIST 1.1. However, there is no prospective randomized study to prove the efficacy and safety of HAIC combined with apatinib and camrelizumab. So this study was designed to evaluate the efficacy and safety of hepatic arterial infusion chemotherapy combined with Apatinib and Camrelizumab versus Apatinib and Camrelizumab to provide a more effective and toxic-tolerable treatment for patients in C-staged Hepatocellular Carcinoma in BCLC classification.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily joins the study and signs an informed consent;
2. Age ≥ 18 years old,both men and women;
3. Clinical or pathologically confirmed unresectable BCLC C-stage hepatocellular carcinoma according to AASLD: HCC with vascular invasion and/or extrahepatic metastasis which is not suitable for radical surgery and/or local therapy, or progressed after surgery and/or local therapy
4. No prior systemic therapy;
5. At least one intrahepatic evaluable tumor existed according to RECIST 1.1;
6. Child-Pugh score small or equal to 6 points ;
7. Patient can swallow tablet normally;
8. ECOG score: 0 to 1 (according to the ECOG score classification);
9. The expected survival is longer than 12 weeks;
10. The laboratory parameters meets the following requirements (no blood components and cell growth factors are allowed within 14 days before the first dose):

    * Absolute neutrophil count ≥ 3.0 × 10^9 / L;
    * Platelets ≥ 80 × 10^9 / L;
    * Hemoglobin ≥ 90 g / L;
    * serum albumin ≥ 28 g / L;
    * Thyroid stimulating hormone (TSH) ≤ 1 × ULN (if abnormalities should be considered at the same time FT3, FT4 levels, patients with FT3 and FT4 levels in normal range can also be enrolled);
    * bilirubin ≤ 1.5 × ULN (within 7 days prior to the first dose);
    * ALT ≤ 3 x ULN and AST ≤ 3 x ULN (within 7 days prior to the first dose);
    * AKP ≤ 2.5 × ULN; serum creatinine ≤ 1.5 × ULN;
11. Patients with active hepatitis B virus (HBV) infection recieve anti-HBV therapy at the screening stage and are willing to receive antiviral therapy throughout the study period; hepatitis C virus (HCV) ribonucleic acid (RNA)-positive patients must receive antiviral therapy according to local standard treatment guidelines;
12. For female that non-surgical sterilization or in childbearing age need to use a medically approved contraceptive (such as an intrauterine device, contraceptive or condom) during the study period and within 3 months after the end of the study treatment period; For female that non-surgical sterilization or in childbearing age must have a negative serum or urine HCG test within 72 hours prior to study enrollment; and must be non-lactating; for male patients whose partner in a childbearing age, effective methods of contraception should be given during the trial and at the end of Camrelizumab injection.

Exclusion Criteria:

1. The patient has any active auto-immune disease or a history of auto-immune disease (such as the following, but not limited to: auto-immune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, thyroid hyperfunction; patients with vitiligo. For patient with history of asthma, complete remission of asthma in childhood without any intervention after adulthood can be included, while those asthma patients who require bronchodilators for medical intervention cannot be included.);
2. The patient is using immunosuppressive agents or systemic hormonal therapy for immunosuppression purposes (dose > 10 mg/day of prednisone or other therapeutic hormones) and continues to be used within 2 weeks prior to enrollment;
3. Severe allergic reactions to other monoclonal antibodies;
4. Known for a history of central nervous system metastasis or hepatic encephalopathy;
5. Having a history of organ transplantation;
6. Patients with clinically symptomatic ascites who require puncture, drainage, or ascites drainage within 3 months, except for those who have a small amount of ascites but no clinical symptoms;
7. Suffering from hypertension, and cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥ 140mmHg or diastolic blood pressure ≥90 mmHg);
8. Suffering heart diseases with clinical symptoms or those not well controlled, such as: (1) heart failure in NYHA class 2 or higher; (2) unstable angina; (3) myocardial infarction occurred within 1 year; (4) clinically symptomatic supraventricular or ventricular arrhythmia requiring treatment or intervention; (5) Tc > 450ms (male); QTc > 470ms (female);
9. Coagulation dysfunction (INR>2.0, PT>16s), bleeding tendency or receiving thrombolysis or anticoagulant therapy, allowing prophylactic use of low-dose aspirin or low molecular heparin;
10. There are significant clinically significant bleeding symptoms or clear bleeding tendency within 3 months before enrollment, such as hemoptysis of 2.5ml or more per day, gastrointestinal bleeding, esophageal varices with bleeding risk, hemorrhagic gastric ulcer or vasculitis, etc. If the fecal occult blood is positive in the baseline period, it can be watched, then gastroscope is needed for those fecal occult blood is still positive. If the gastroscope indicates severe esophageal varices, it cannot be enrolled, except for those who have undergone gastroscopy within a month or less to exclude such cases);
11. Events of arterial/venous thrombosis occurring within the first 6 months of enrollment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
12. There are known hereditary or acquired bleeding and thrombophilia (such as hemophilia patients, coagulopathy, thrombocytopenia, etc.);
13. Urine routine indicates that urine protein ≥ ++ and 24-hour urine protein amount > 1.0g was confirmed;
14. The patient has active infection, unexplained fever (≥38.5 °C) within 3 days before administration, or baseline white blood cell count>15×109/L; 15 Patients with congenital or acquired immunodeficiency (such as HIV-infected patients);

16. HBV-DNA>2000 IU/ml (or 104 copies/ml); or HCV-RNA>103 copies/ml; or HBsAg+ and anti-HCV antibody positive patients; 17. The patient has had other malignant tumors in the past 3 years or at the same time (except for cured skin basal cell carcinoma and cervical carcinoma in situ); 18. Patients with bone metastases who had received palliative radiotherapy >4% of the bone marrow area within 4 weeks prior to participation in the study; 19. Patients have previously received other anti-PD-1 antibody therapy or other immunotherapy against PD-1/PD-L1, or have received apatinib before; 20. Inoculation of a live vaccine within less than 4 weeks prior to study or possibly during the study period; 21. Pregnant or lactating women, or women of childbearing age who are unwilling to take contraceptive measures; 22. According to the investigators, the patient has other factors that may affect the results of the study or lead to the termination of the study, such as alcohol abuse, drug abuse, other serious diseases (including mental illness) requiring combined treatment, and serious laboratory tests, abnormalities, accompanied by factors such as family or society, which may affect the safety of enrolled patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The progression-free survival (PFS) by RECIST 1.1 | From date of first dose of study drug to the date of first documentation of disease progression or death, whichever occurs first (up to approximately 3 years)

SECONDARY OUTCOMES:
The progression-free survival (PFS) by mRECIST | From date of first dose of study drug to the date of first documentation of disease progression or death, whichever occurs first (up to approximately 3 years)
The overall survival (OS) | From date of first dose of study drug to the date of first documentation of death from any cause, whichever occurs first (up to approximately 3 years)
Time to progress (TTP) by RECIST 1.1 and mRECIST | From date of first dose of study drug until disease progression or death (up to approximately 3 years)
Time to response (TTR) by RECIST 1.1 and mRECIST | From date of first dose of study drug until the first documentation of CR or PR
Duration of response (DOR) by RECIST 1.1 and mRECIST | From the first documentation of CR or PR to the first date of documentation of disease progression or death whichever occurs first (up to approximately 3 years)
  DOR is defined as the time from the first documentation of CR or PR to the date of first documentation of disease progression or death (whichever occurs first) as assessed by RECIST 1.1 and mRECIST
Objective response rate (ORR) by RECIST 1.1 and mRECIST | From date of first dose of study drug until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to approximately 3 years)
  ORR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) at the time of data cutoff as assessed by RECIST 1.1 and mRECIST
The disease control rate (DCR) | From date of first dose of study drug until disease progression, stable disease, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to approximately 3 years)
  DCR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) or stable disease (SD) at the time of data cutoff as assessed by RECIST 1.1 and mRECIST
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From the start date of the Treatment Phase until date of death from any cause (up to approximately 3 years)

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-Sen University, Guanzhou, Guangdong
  - Xiangya Hospital of Central South University, Changsha, Hunan

REFERENCES:
- [Background] Lyu N, Kong Y, Mu L, Lin Y, Li J, Liu Y, Zhang Z, Zheng L, Deng H, Li S, Xie Q, Guo R, Shi M, Xu L, Cai X, Wu P, Zhao M. Hepatic arterial infusion of oxaliplatin plus fluorouracil/leucovorin vs. sorafenib for advanced hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):60-69. doi: 10.1016/j.jhep.2018.02.008. Epub 2018 Feb 20. PMID 29471013
- [Background] He M, Li Q, Zou R, Shen J, Fang W, Tan G, Zhou Y, Wu X, Xu L, Wei W, Le Y, Zhou Z, Zhao M, Guo Y, Guo R, Chen M, Shi M. Sorafenib Plus Hepatic Arterial Infusion of Oxaliplatin, Fluorouracil, and Leucovorin vs Sorafenib Alone for Hepatocellular Carcinoma With Portal Vein Invasion: A Randomized Clinical Trial. JAMA Oncol. 2019 Jul 1;5(7):953-960. doi: 10.1001/jamaoncol.2019.0250. PMID 31070690